CLINICAL TRIAL: NCT00568074
Title: Efficacy and Safety of Repaglinide, Glurenorm® and Glucobay® in Chinese Subjects With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of Repaglinide, Glurenorm® and Glucobay® in Chinese Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGEE-1555
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide; gliquidone; Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: repaglinide
Drug: Glurenorm®
Drug: Glucobay®

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to compare the efficacy and safety of repaglinide and Glurenorm® and Glucobay® given as the mono-therapy in Chinese subjects being treatment-naive type 2 diabetics.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* No previous treatment for diabetes
* HbA1c: 7.0-12.0%

Exclusion Criteria:

* Type 1 diabetes
* Uncontrolled treated/untreated hypertension
* Any condition that the Investigator and/or Sponsor feels would interfere with trial participation or evaluation of results
* Pregnancy, breast-feeding, the intention of becoming pregnant or judged to be using inadequate contraceptive measures (adequate contraceptive measures are: sterilisation, intra-uterine device (IUD), oral contraceptives or barrier methods)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2003-12-16; Primary Completion 2004-09-02 (Actual); Study Completion 2004-09-02 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 3 months of treatment

SECONDARY OUTCOMES:
fasting blood glucose
hypoglycaemia episodes
adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (3):
- China (3):
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality
  - Novo Nordisk Investigational Site, Chengdu, Sichuan
  - Novo Nordisk Investigational Site, Beijing

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com